CLINICAL TRIAL: NCT02416557
Title: Effect of Positive End Expiratory Pressure on Intraoperative Body Temperature in Patients Undergoing Spine Surgery; a Prospective Randomized Study
Brief Title: Effect of PEEP on Intraoperative Hypothermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Intraoperative hypothermia
Record Dates: First submitted 2015-04-06; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Spinal Diseases
MeSH Terms: conditions — Spinal Diseases | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group P (Experimental): Patients using positive end-expiratory pressure (PEEP) of 10 cmH2O (centimeter of water) intraoperatively
  Interventions: Procedure: PEEP
- Group C (No Intervention): Patients using no positive end-expiratory pressure (zero PEEP) intraoperatively

INTERVENTIONS:
Procedure: PEEP — application of 10 cmH2O (centimeter of water) positive end expiratory pressure during mechanical ventilation
  Other Names: positive end expiratory pressure
  Arms: Group P

SUMMARY:
Intraoperative hypothermia is associated with many clinical adverse outcomes. Many techniques were applied to prevent intraoperative hypothermia, and positive end-expiratory pressure (PEEP) has been known to blunt intraoperative hypothermia by increasing thermoregulatory vasoconstriction threshold. The investigators assessed the effect of PEEP on the prevention of intraoperative hypothermia during spine surgery in prone position.

DETAILED DESCRIPTION:
It is well known that intraoperative hypothermia is associated with postoperative adverse clinical outcomes in various study populations. Intraoperative hypothermia has various adverse effects including impaired drug clearance, cold diuresis and hypovolemia, immunosuppression with increased infection risk, electrolyte disorders, coagulopathy with impaired platelet function, negative nitrogen balance, shivering, insulin resistance, and myocardial events. Numerous methods have been introduced to prevent intraoperative hypothermia, such as warming of infusion fluid, forced-air warming, heat-pads, heated water mattress, and heated humidifiers. However, in patients undergoing lumbar spine surgery in the prone position, these methods to prevent intraoperative hypothermia may partially effective because these methods, in clinical practice, have a significant limitation in their application.

Positive end-expiratory pressure (PEEP) reduces the venous return by increasing intrathoracic pressure. This causes carotid unloading, which leads to a secondary peripheral vasoconstriction by increasing thermoregulatory vasoconstriction threshold and blunts intraoperative hypothermia. Previous studies demonstrated that intraoperative PEEP significantly attenuated the extent of intraoperative hypothermia in patients undergoing tympanoplasty. However, the beneficial effect of PEEP on thermoregulation is not investigated in patients with the prone position for spinal surgery.

The investigators hypothesized that PEEP can reduce the extent of intraoperative hypothermia via thermoregulatory modulation. In this study, the investigators investigated the effect of PEEP on intraoperative core body temperature and the incidence of intraoperative hypothermia in patients undergoing spinal surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for elective spine surgery requiring more than 3 hours

Exclusion Criteria:

* Patients who do not agree to the study
* Patients with or American Society of Anesthesiologists (ASA) physical status class 3 or more
* Patients with thyroid disease, peripheral vascular diseases, uncontrolled diabetes or hypertension
* Patients with morbid obesity (BMI >35 kg/m2)
* Patients with clinically severe pulmonary disease
* Patients undergoing simultaneous anterior and posterior lumbar fusion surgery were also excluded.
* Patients with taking non-steroidal anti-inflammatory drug within two weeks
* Patients with preoperative fever or hypothermia
* Patients with intraoperative intentional hypothermia for neuroprotection

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Body temperature as assessed by esophageal temperature probe | 180 minutes after the completion of anesthesia induction
  Body temperature is assessed by esophageal temperature probe. The investigators used body temperature at 180 minutes after anesthesia induction as a primary outcome

SECONDARY OUTCOMES:
Thermoregulatory vasoconstriction threshold | until 180 minutes after the completion of anesthesia induction
  The time of the difference in skin temperature between forearm and fingertip becoming zero.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea

REFERENCES:
- [Background] Yamasaki H, Tanaka K, Funai Y, Suehiro K, Ikenaga K, Mori T, Osugi H, Nishikawa K. The impact of intraoperative hypothermia on early postoperative adverse events after radical esophagectomy for cancer: a retrospective cohort study. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):943-7. doi: 10.1053/j.jvca.2014.02.013. PMID 25107714
- [Background] Nakajima Y, Mizobe T, Takamata A, Tanaka Y. Baroreflex modulation of peripheral vasoconstriction during progressive hypothermia in anesthetized humans. Am J Physiol Regul Integr Comp Physiol. 2000 Oct;279(4):R1430-6. doi: 10.1152/ajpregu.2000.279.4.R1430. PMID 11004013
- [Background] Jung KT, Kim SH, Lee HY, Jung JD, Yu BS, Lim KJ, So KY, Lee JY, An TH. Effect on thermoregulatory responses in patients undergoing a tympanoplasty in accordance to the anesthetic techniques during PEEP: a comparison between inhalation anesthesia with desflurane and TIVA. Korean J Anesthesiol. 2014 Jul;67(1):32-7. doi: 10.4097/kjae.2014.67.1.32. Epub 2014 Jul 29. PMID 25097736